CLINICAL TRIAL: NCT06070584
Title: Effect of Respiratory Muscle Training on Lung Function on Quarry Workers in Minia Government Egypt
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4/23
Record Dates: First submitted 2023-09-24; First posted 2023-10-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Lung Function Decreased
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): received aerobic exercises only
  Interventions: Procedure: aerobic exercises with electrical treadmill for 30 min and inspiratory muscle training for 10 minutes.,
- Group B (Experimental): aerobic exercises with moderate intensity in the form of walking on electrical treadmill
  Interventions: Procedure: aerobic exercises with electrical treadmill for 30 min and inspiratory muscle training for 10 minutes.,

INTERVENTIONS:
Procedure: aerobic exercises with electrical treadmill for 30 min and inspiratory muscle training for 10 minutes., — aerobic exercises with moderate intensity in the form of walking on electrical treadmill

SUMMARY:
forty quarry workers participated in the study with age range (40-60 years), body mass index (BMI) from 25 to 34.9 kg/m2 (over weight and class 1 obesity). The patients divided into two groups randomly. (Group A) received aerobic exercises (Group B) receive aerobic exercises with moderate intensity in the form of walking on electrical treadmill for 30 min and inspiratory muscle training for 10 minutes., 3 sessions per week for 8 consecutive weeks. Pulmonary function test was applied by spirometry to assess lung function

ELIGIBILITY:
Inclusion Criteria:

* quarry workers working in the quarries for five years ago at least saver from chest diseases\\
* BMI ranged from 25 to 34.9 kg/cm2

Exclusion Criteria:

* Subject with infected chest disease, unstable mental condition and chest cancer patients
* musculoskeletal disease

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
adequate lung function | 8 weeks
  Spirometer test, The patient was instructed to take a big breath in and then exhale as forcefully and quickly as they could, continuing until there was no more air remaining, in order to measure FVC and FEV1
patient satisfaction | 8 weeks
  VAS scoring, (no pain=0) and the other end (worst pain=10).

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No